CLINICAL TRIAL: NCT03452124
Title: The Effects of I Quit Ordinary Smoking on the Arterial Wall and Endothelial Glycocalyx Properties of Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate Professor, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IQOS-ATTIKON
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQOS (Active Comparator): I quit ordinary smoking (IQOS) assistes cessation program
  Interventions: Device: I quit ordinary smoking (IQOS)
- Smoker control (Active Comparator): Conventional cigarette smoking continuation
  Interventions: Other: Conventional cigarette

INTERVENTIONS:
Device: I quit ordinary smoking (IQOS) — I quit ordinary smoking (IQOS) assisted cessation program
  Arms: IQOS
Other: Conventional cigarette — Conventional cigarette smoking continuation
  Arms: Smoker control

SUMMARY:
I quit ordinary smoking (IQOS) is proposed as a bridge to smoking cessation. In this study the investigators will examine its effects on aortic elasticity, glycocalyx integrity, and exhaled carbon monoxide (CO) concentration, both acutely and after 1 month of use.

DETAILED DESCRIPTION:
Two smokers groups matched for age and sex will be assessed:

1. a group of 30 current smokers with no diagnosed cardiovascular disease as the control group for chronic phase
2. a group of 30 current smokers with no diagnosed cardiovascular disease who will be using the I quit ordinary smoking (IQOS) for 1 month.

In the acute phase all 60 smokers will undergo a "sham" smoking for 7 minutes. Afterwards all 60 smokers will be randomized to smoke either a normal cigarette or IQOS and the after 60 minute washout period these subjects will be crossed over to the altenate mode of smoking (IQOS or normal cigarette respectively).

After the completion of the acute phase all 60 smokers will start the use of IQOS for one month.

In the acute phase, measurements will be performed at baseline, after sham smoking and after smoking of the normal cigarette or IQOS. The chronic phase measurements will be performed 1 month after use IQOS. Thirty current smokers of similar age and sex will serve as controls and will have measurements at baseline and 1 month after baseline assessment.

In both phases the investigators will assess: a) the aortic pulse wave velocity (PWV) and augmentation index (AIx) by Arteriograph and Complior; b) the perfusion boundary region of the sublingual arterial microvessels using Sideview, Darkfield imaging (Microscan, Glycocheck); c) the exhaled carbon monoxide (CO) level (parts per million -ppm) as a smoking status marker; d) the vital signs; e) an electrocardiogram; and f) plasma levels of C- reactive protein (CRP), transforming growth factor-b (TGF-b), lipoprotein associated phospholipase A2 (LP- LPA2), tumor necrosis factor- α (TNF-α), interleukins 6 and 10 (IL-6 and -10), procollagen propeptide type III (PIIINP), matrix metalloproteinase 2 and 9 (MMP-2 and -9), and macrophage-colony stimulating factor (MCSF), malondialdehyde (MDA) and protein carbonyls (PCs).

ELIGIBILITY:
Inclusion Criteria:

* Active conventional cigarette smoker

Exclusion Criteria:

* Health condition adversely affected by smoking
* History or presence of cardiovascular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute I quit ordinary smoking (IQOS) effects on pulse wave velocity | 7 minutes
  Acute I quit ordinary smoking (IQOS) effects on pulse wave velocity (PWV, m/s) using tonometry
Acute I quit ordinary smoking (IQOS) effects on Exhaled Carbon monoxide (CO) | 7 minutes
  CO concentration was measured the exhaled carbon as parts per million-ppm by the device Smokerlyzer, Covita, Bedfont, CA, USA). Participants were instructed not to smoke the night before and the morning before the CO measurements and to hold their breath for 10 sec before exhaling to the mouthpiece.
Acute I quit ordinary smoking (IQOS) effects on endothelial glycocalyx thickness | 7 minutes
  Acute I quit ordinary smoking (IQOS) effects on endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublinqual arterial microvessels
Chronic I quit ordinary smoking (IQOS) effects on pulse wave velocity | 1 month
  Chronic I quit ordinary smoking (IQOS) effects on pulse wave velocity (PWV, m/s) using tonometry
Chronic I quit ordinary smoking (IQOS) effects on endothelial glycocalyx thickness | 1 month
  Chronic I quit ordinary smoking (IQOS) effects on endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublinqual arterial microvessels
Chronic I quit ordinary smoking (IQOS) effects in left ventricular function | 1 month
  Left Ventricular function is assessed by Global Longitudinal Strain by speckle tracking echocardiography
Chronic I quit ordinary smoking (IQOS) effects on endothelial function | 1 month
  Endothelial function was assessed by measuring coronary flow reserve of Left anterior descending artery. Coronary flow reserve was estimated by Doppler echocardiography as the ratio of coranary flow velocity after bolus intravenous adenosine infusion to coronary flow velocity at rest.
Chronic I quit ordinary smoking (IQOS) effects on endothelial function | 1 month
  Endothelial function was assessed by measuring Flow Mediated Vasodilation (FMD) using sonography. During a FMD test, vasodilation occurs following an acute increase in blood flow, typically induced via circulatory arrest in the arm (supra-systolic cuff occlusion) for a period of time. FMD is the percent of increase in brachial artery diameter after occlusion.
Chronic I quit ordinary smoking (IQOS) effects on Exhaled Carbon monoxide (CO) | 1 month
  CO concentration was measured the exhaled carbon as parts per million-ppm by the device Smokerlyzer, Covita, Bedfont, CA, USA). Participants were instructed not to smoke the night before and the morning before the CO measurements and to hold their breath for 10 sec before exhaling to the mouthpiece.

SECONDARY OUTCOMES:
Acute I quit ordinary smoking (IQOS) effects on platelet activation. | 7 minutes
  Platelet activation was estimated by measuring blood levels of Thromboxane B2 (Thromboxane B2 EIA Kit Cayman Ann Arbor MI USA) A commercially available ELISA kit was used with an assay range 1.6-1000 pg/ml.
Chronic I quit ordinary smoking (IQOS) effects on myocardial work. | 1 month
  Myocardial work (MW) was estimated by combining echo-derived left ventricular (LV) strain with brachial blood pressure to construct LV strain-pressure curves non-invasively. Brachial cuff systolic pressure measurements provide the peak systolic LV pressure value, which is combined with the input of valvular timing events that define isovolumetric and ejection phases, allowing the construction of an LV-pressure curve. This is combined with LV strain data into a pressure-strain loop (PSL), the area within which represents MW. Global MW index (GWI) is defined as the work within the LV PSL from mitral valve closure to mitral valve opening, while constructive MW (GCW) is the component of MW that contributes to LV ejection. On the contrary, wasted MW (GWW) is the work wasted as myocyte lengthening during systole, which does not contribute to LV ejection. MW efficiency (GWE) is defined as the ratio of GCW to the sum of GCW and GWW [GWE= GCW/ (GCW+GWW)].
Chronic I quit ordinary smoking (IQOS) effects on arterial stiffness. | 1 month
  Arterial stiffness was estimated by calculating Total arterial compliance (TAC). TAC was evaluated utilising the stroke volume (SV) to pulse pressure (PP) ratio (SV/PP), based on the two-element Windkessel model; SV measurements were derived from two-dimensional echocardiography.
Chronic I quit ordinary smoking (IQOS) effects on platelet activation. | 1 month
  Platelet activation was estimated by measuring blood levels of Thromboxane B2 (Thromboxane B2 EIA Kit Cayman Ann Arbor MI USA) A commercially available ELISA kit was used with an assay range 1.6-1000 pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — Attikon University General Hospital
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Ikonomidis I, Vlastos D, Kostelli G, Kourea K, Katogiannis K, Tsoumani M, Parissis J, Andreadou I, Alexopoulos D. Differential effects of heat-not-burn and conventional cigarettes on coronary flow, myocardial and vascular function. Sci Rep. 2021 Jun 3;11(1):11808. doi: 10.1038/s41598-021-91245-9. PMID 34083663